CLINICAL TRIAL: NCT03828565
Title: Decrease of Post-operative Complications by SCVO2 Monitoring an Optimisation of Cardiac Flow : Multicentric Randomized Control in Single Blind Study
Brief Title: Decrease of Post-operative Complications by SCVO2 Monitoring an Optimisation of Cardiac Flow
Acronym: OCOSO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-37; IDRCB (Other: 2018-A02511-54)
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Flow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ScvO2 group (Active Comparator): ScvO2 and Pulse Pressure Variation (PPV) : every 30 min (%) ScvO2 Evolution in case of corrective maneuver (%) PPV evolution in case of filling test (%)
  Interventions: Procedure: ScvO2 Perioperative continue monitoring
- Control group (No Intervention): End-systolic Volume (ESV) : every 30 min (mL) ESV evolution in case of filling test (%)

INTERVENTIONS:
Procedure: ScvO2 Perioperative continue monitoring — ScvO2 Perioperative continue monitoring with PreSep® system. If SvcO2 is less than 65% or decreases by more than 10% of its base value, the other parameters affecting ScvO2 (BIS (40-60% objective), Hb (objective> 8g / dL), SaO2 (objective> 94%)) are evaluated. If, after correcting for these parameters, the ScvO2 is not corrected, the preload-dependence parameters are evaluated (variation of the pulsed pressure) to guide the vascular filling: VF of 250 mL of crystalloids if PPV> 13%, norepinephrine if PPV<9%, reassess if PPV between 9 and 13%.
  If VF or norepinephrine does not correct ScvO2 (> 65%), a measurement of arterial lactate is performed. If lactatemia is> 2 mmol / L, a positive inotrop is introduced after ETO if possible. If lactatemia is <2 mmol / L, a return to the evaluation phase of the parameters influencing ScvO2 is necessary.
  Arms: ScvO2 group

SUMMARY:
In operating theater, one of the bigger purpose of anesthetist-resuscitator is to optimize vascular filling (VF) because of a failure or an excess of filling is deleterious for the patient. Several studies have assessed the traditionnal VF based on the clinic and the VF guided by quantitative critereas. Thus studies have showed a decrease of morbidity and duration of patients' stay whose the VF was guided even on the long term. So, formal recommandations of experts (FRE) on the perioperative filling strategy of the SFAR ( Anesthesia and Resuscitation Francophone Society) advise to titrate the perioperative vascular filling of high risk patients guiding on a mesure of end-systolic volume (ESV). The inscrease of ESV answering to filling confirmed the VF realized is relevant and authorized its pursuite while the absence of an increase of the ESV after a filling test signifies the useless and deleterious character of this one. The optimization of perioperative hemodynamics consists in adapting the patient's cardiac output to his metabolic needs. ETO, Swan-Ganz: limit of its application to the routine. The central venous oxygen saturation (ScvO2) is simple and safe, the evaluation of the adjustment of O2 inputs compared to the needs. The industry has developed continuous monitoring systems by reflection spectrophotometry using optical fibers installed in the central venous pathways. In daily practice, the stricto sensu application of FRE leads to administering an VF up to the limit of the preload dependence without evaluating the adequacy of the cardiac output, which is not a physiological situation. This filling is therefore sometimes performed solely on the criteria of preload dependence while it is potentially deleterious for the patient. No study has compared a strategy based on the use of ScvO2 and preload dependence with current recommendations based solely on preload dependence. Our hypothesis is that the continuous monitoring of the ScvO2 in the superior cave territory in intraoperative would allow to detect the patients with an inadequacy of the cardiac output and thus to select the only ones requiring a vascular filling. This would reduce postoperative complications related to overfilling, without exposing the patient to episodes of tissue hypoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* >50 years old
* ASA score ≥ 2
* requiring a major intra-abdominal scheduled surgery
* lasting more than 90 min
* in the visceral surgery, vascular surgery, urological surgery and gynecological surgery sectors

Exclusion Criteria:

* <18 years old
* Pregnant or brest feeding patients
* no consentement
* Unstable acute pathology at the time of surgery (acute heart, respiratory or renal failure, severe sepsis or septic shock, hemorrhagic shock);
* rhythm disorders type ACFA early intervention;
* Palliative surgery, ASA 5;
* Patient under guardianship or curatorship.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Difference of the CCI score at day 5 between patients of ScvO2 group and patient of control group. | Day 5
  CCI score : Comprehensive Complication Index. Allow to integrate all the postoperative complications and their respectives severities. From 0 (No complication) to 100 (death of the patient)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier Arnaud, Study Director — APHM
Locations (1):
- Laurent Zieleskiewicz, Marseille, PACA, France

REFERENCES:
- [Derived] Pastene B, Bernat M, Baumstark K, Bezulier K, Gricourt Y, De Guibert JM, Charvet A, Colin M, Leone M, Zieleskiewicz L. OCOSO2: study protocol for a single-blinded, multicentre, randomised controlled trial assessing a central venous oxygen saturation-based goal-directed therapy to reduce postoperative complications in high-risk patients after elective major surgery. Trials. 2023 Oct 11;24(1):659. doi: 10.1186/s13063-023-07689-z. PMID 37821968